CLINICAL TRIAL: NCT01353131
Title: Personalized Risk Identification and Management for Arrhythmias and Heart Failure by 12 Lead Electrocardiogram and Cardiac Magnetic Resonance Imaging.
Brief Title: Personalized Risk Identification and Management for Arrhythmias and Heart Failure by ECG and MRI
Acronym: PRIMERI
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00031964
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Inpatients and Outpatients With Routine 12-lead ECG
Keywords: electrocardiogram; cardiac magnetic resonance; heart failure; sudden cardiac death; ECG scoring; Delayed enhancement
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ECG Screening: 1000 patients with moderate to high risk determined by stratification algorithm based on the electronic analysis of 69,088 routine 12-lead ECGs performed in a large medical institution during a 6 month period by combining previously established indices of abnormal repolarization (wide QRS-T angle) with validated measures of myocardial damage (Selvester QRS score) excluding those > 70 years of age or with LV ejection fraction ≤ 35%, or at a high risk of dying within 3 years from cancer, end stage cardiac, pulmonary, renal, immunologic or neurologic diseases excluded on clinical data obtained through medical record.

SUMMARY:
Prevention of myocardial functional deterioration and sudden cardiac death among individuals of intermediate risk remains one of the most elusive frontiers of contemporary medicine. While most of these individuals are known to have had contact with the medical system, they are frequently not considered to be at high risk until far advanced along one or multiple disease processes leading to irreversible myocardial loss and electric instability. The goal of this proposal is to determine the prognostic power of combining specific measures of ventricular architecture, myocardial structure and electrical function for the early identification of individuals at risk to develop ventricular arrhythmias and progressive myocardial failure leading to severe cardiovascular outcomes and death.

DETAILED DESCRIPTION:
During C-TRIP Stage 1 we refined a risk stratification algorithm based on the electronic analysis of 69,088 routine 12-lead ECGs performed in a large medical institution during a 6 month period by combining previously established indices of abnormal repolarization (wide QRS-T angle) with validated measures of myocardial damage (Selvester QRS score). Among patients considered at risk, 4.9% had perished 18 months later and among the survivors those > 70 years of age or with LV ejection fraction ≤ 35%, or at a high risk of dying within 3 years from cancer, end stage cardiac, pulmonary, renal, immunologic or neurologic diseases, were excluded using a simple and reproducible screening arborescence based on the digital medical record. From the pool of remaining at risk patients derived from the application of the same screening methods in three other similarly large academic institutions, a sample of 1100 individuals will be recruited for further risk stratification as participants of the C-TRIP Stage 2 prospective study. For C-TRIP Stage 2, patients will undergo detailed phenotypic studies including contrast-enhanced cardiac MRI, ECG Holter recordings at rest and during a 6 minute walk, signal averaged ECG and biomarkers of inflammation, myocardial ischemia and stress, as well as indices of collagen synthesis and turnover. Patients will be followed for 3 years for the development of a combined clinical outcome including mortality (all cause, cardiac and sudden cardiac death) and hospitalization for non-fatal myocardial infarction, acute coronary syndromes, ventricular arrhythmias and heart failure. From the combination of selected phenotypic markers of poor outcome, a risk score will be developed and used for the design of prophylactic strategies aimed at curbing premature sudden cardiac death and end-stage cardiac disease among patients currently classified as having intermediate levels of risk.

ELIGIBILITY:
Inclusion Criteria:

* general hospital population with routine 12-lead ECG with abnormal repolarization (wide QRS-T angle>100°) with validated measures of myocardial damage (Selvester QRS score>5)

Exclusion Criteria:

* LVEF <35%
* age>70 years
* eGFR<45mL/min
* no ICD or PM
* no high risk of dying within 3 years from cancer, end stage cardiac, pulmonary, immunologic or neurologic diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We refined a risk stratification algorithm based on the electronic analysis of 69,088 routine 12-lead ECGs performed in a large medical institution during a 6 month period by combining previously established indices of abnormal repolarization (wide QRS-T angle) with validated measures of myocardial damage (Selvester QRS score).
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2010-05; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joao AC Lima, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Division of Cardiology, Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Mewton N, Strauss DG, Rizzi P, Verrier RL, Liu CY, Tereshchenko LG, Nearing B, Volpe GJ, Marchlinski FE, Moxley J, Killian T, Wu KC, Spooner P, Lima JA. Screening for Cardiac Magnetic Resonance Scar Features by 12-Lead ECG, in Patients with Preserved Ejection Fraction. Ann Noninvasive Electrocardiol. 2016 Jan;21(1):49-59. doi: 10.1111/anec.12264. PMID 26806840
- [Derived] Murthy S, Rizzi P, Mewton N, Strauss DG, Liu CY, Volpe GJ, Marchlinski FE, Spooner P, Berger RD, Kellman P, Lima JA, Tereshchenko LG. Number of P-wave fragmentations on P-SAECG correlates with infiltrated atrial fat. Ann Noninvasive Electrocardiol. 2014 Mar;19(2):114-21. doi: 10.1111/anec.12084. Epub 2013 Sep 9. PMID 24620844
- [Derived] Tereshchenko LG, Rizzi P, Mewton N, Volpe GJ, Murthy S, Strauss DG, Liu CY, Marchlinski FE, Spooner P, Berger RD, Kellman P, Lima JA. Infiltrated atrial fat characterizes underlying atrial fibrillation substrate in patients at risk as defined by the ARIC atrial fibrillation risk score. Int J Cardiol. 2014 Mar 1;172(1):196-201. doi: 10.1016/j.ijcard.2014.01.012. Epub 2014 Jan 22. PMID 24485635